CLINICAL TRIAL: NCT03635151
Title: Caregiver Self-Management Needs Through Skill-Building
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Tamilyn Bakas, Professor and Jane E. Procter Endowed Chair, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-8508; 1R21NR016992-01A1 (NIH)
Record Dates: First submitted 2018-07-24; First posted 2018-08-17 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Family Caregivers; Stroke
Keywords: Clinical trial
MeSH Terms: conditions — Stroke | interventions — Population Groups; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TASK III Group (Experimental): The Telephone Assessment and Skill-Building Kit (TASK III) group
  Interventions: Behavioral: Telephone Assessment and Skill-Building Kit (TASK III) Group
- ISR Group (Active Comparator): The Information, Support, and Referral (ISR) group
  Interventions: Behavioral: Information Support and Referral (ISR) Group

INTERVENTIONS:
Behavioral: Telephone Assessment and Skill-Building Kit (TASK III) Group — The TASK III group will receive a TASK III Resource Guide that we developed and 8 weekly calls from a nurse. The nurse will call again a month later. The TASK III nurse will help you assess your needs and concerns, build your skills as a caregiver, and refer you to community resources.
  Arms: TASK III Group
Behavioral: Information Support and Referral (ISR) Group — The ISR group will receive an American Heart Association brochure and 8 weekly calls from a nurse. The nurse will call again a month later. The ISR nurse will provide information, support, and referral to community resources.
  Arms: ISR Group

SUMMARY:
Caring for a family member after a stroke can be very difficult and worsen the physical and mental health of untrained caregivers. The Telephone Assessment and Skill-Building Kit (TASK III) intervention is a unique, comprehensive caregiver intervention program that enables caregivers to develop the necessary skills to manage care for the survivor, while also taking care of themselves. The long-term goal of this study is to offer training and support for family caregivers through an efficacious, cost-effective program.

DETAILED DESCRIPTION:
Stroke is a leading cause of serious, long-term disability, and has a very sudden onset; families are often thrust into providing care without any training from health care providers. Studies have shown that caregiving without training can be detrimental to caregiver's physical and mental health, which can impede survivor rehabilitation and lead to institutionalization and higher societal costs. Unlike existing stroke caregiver interventions that require costly face to face interactions, and that focus primarily on the survivor's care, the Telephone Assessment and Skill-Building Kit (TASK II) is delivered completely by telephone, and empowers caregivers to address both their own and the survivor's needs using innovative skill-building strategies. Aligned with current patient and caregiver guidelines, TASK II has demonstrated evidence of content validity, treatment fidelity, caregiver satisfaction, and efficacy for reducing depressive symptoms; however, future development of TASK II requires a stronger focus on self-management strategies to improve caregiver health, and enhanced use of other telehealth modes of delivery prior to implementation into ongoing stroke systems of care. The purpose of this study is to optimize the TASK III intervention through the innovative leveraging of technologies and theoretically-based self-management strategies to improve caregiver health. Specific Aim 1 consists of focus groups and individual interviews with 40 experts (10 interdisciplinary researchers, 10 technology experts, 10 clinicians and clinical leaders, and 10 stroke family caregivers) to provide preferences about essential areas of new self-management content, proposed technologies (e.g., iBook, eBook, interactive website, FaceTime, Zoom), and future implementation strategies to inform a novel TASK III prototype. Specific Aim 2 will determine feasibility of the TASK III intervention with a pilot study of 74 stroke caregivers randomized to TASK III or an Information, Support, and Referral (ISR) group in preparation for a larger randomized controlled clinical trial. Recruitment, retention, treatment fidelity, satisfaction, and technology ratings will be obtained for both TASK III and ISR groups who will receive 8 weekly sessions with a booster session 4 weeks later. Outcome measures will be explored at baseline, 8 weeks (end of intervention), and 12 weeks (after booster). If TASK III is shown to be efficacious in a future randomized controlled clinical trial, our next goal will be to translate TASK III into ongoing stroke systems of care; and, someday to adapt it for use among caregivers with other debilitating/chronic conditions providing a tremendous public health impact.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Primary caregiver (unpaid family member or significant other providing care for a stroke survivor)
* Must be providing care after discharge to the home setting (for Specific Aim 2)
* Fluent in the English language
* Access to telephone or computer
* No difficulties hearing or talking by telephone or computer
* (Specific Aim 1) Willing to participate in an online or telephone focus group or an online or telephone individual interview. Some interviews or focus groups may be offered face to face.
* (Specific Aim 2) Willing to participate in 9 calls from a nurse and 3 data collection interviews.

Exclusion Criteria:

Excluded if the survivor:

* Had not had a stroke
* Did not need help from the caregiver
* Was going to reside in a nursing home or long-term care facility

Excluded if the caregiver:

* Scores <16 on the Oberst Caregiving Burden Scale Task Difficulty Subscale (for Specific Aim 2)
* Scores < 4 on a 6-item cognitive impairment screener.

Excluded if the caregiver or survivor is:

* Prisoner or on house arrest
* Pregnant
* Terminal illness (e.g., late stage cancer, end-of-life condition, renal failure requiring dialysis)
* History of Alzheimer's, dementia, or severe mental illness (e.g., suicidal tendencies, schizophrenia, severe untreated depression or manic depressive disorder)
* History of hospitalization for alcohol or drug abuse

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamilyn Bakas, PhD, RN, Principal Investigator — University of Cincinnati College of Nursing
Locations (1):
- University of Cincinnati College of Nursing, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bakas T, McCarthy MJ, Israel J, Brehm BJ, Dunning K, Rota M, Turner M, Miller EL. Adapting the telephone assessment and skill-building kit to the telehealth technology preferences of stroke family caregivers. Res Nurs Health. 2021 Feb;44(1):81-91. doi: 10.1002/nur.22075. Epub 2020 Oct 19. PMID 33075163
- [Result] Bakas T, Jones H, Israel J, Kum C, Miller EL. Designing and Evaluating a Goal-Setting Tip Sheet for Stroke Family Caregiver Health. Rehabil Nurs. 2021 Sep-Oct 01;46(5):279-288. doi: 10.1097/RNJ.0000000000000306. PMID 33512120
- See also: TASK III Study Website — https://www.task3web.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TASK III Group | ISR Group
Started | 36 | 38
Completed | 31 | 34
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TASK III Group | ISR Group | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 56 (17) | 57 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 34 | 38 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 25 | 27 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Patient Health Questionnaire Depression Scale (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — Depressive symptoms measured by the Patient Health Questionnaire Depression Scale (PHQ-9). Caregiver depressive symptoms are measured by the Patient Health Questionnaire Depression Scale (PHQ-9) consisting of 9 items rated on a response scale ranging from 0 = Not at all to 3 = Nearly every day. Items are summed for a total score with a possible range of 0 to 27. Higher scores indicate higher depressive symptoms.
  units on a scale | 5.36 (6.02) | 4.95 (3.88) | 5.15 (5.01)
Bakas Caregiving Outcomes Scale (BCOS) [Mean (Standard Deviation); unit: units on a scale] — Caregiver life changes (i.e., changes in social functioning, subjective well-being, and physical health as a result of providing care) are measured by the Bakas Caregiving Outcomes Scale (BCOS). The BCOS consists of 15 items rated on a response scale ranging from -3 (changed for the worst) to +3 (Changed for the best). The items are recoded (-3= 1) (-2 = 2) (-1 = 3) (0 = 4) (1 = 5) (2 = 6) (3 = 7). The recoded responses to the 15 items are summed for a total score with a possible range of 15-105. Higher scores indicate more positive life changes as a result of providing care.
  units on a scale | 51.72 (9.71) | 53.71 (12.95) | 52.74 (11.45)
Unhealthy Days [Mean (Standard Deviation); unit: Days] — Caregiver unhealthy days are measured using the Unhealthy Days (UD) measure consisting of two items: How many days during the past 30 days was your physical health not good?; How many days during the past 30 days was your mental health not good? These items range from 0 = no unhealthy days to 30 = 30 unhealthy days. The two items are summed for a total score, with a cap of 30 days. Higher scores indicate more unhealthy days in the past 30 days.
  Days | 9.03 (10.57) | 9.97 (9.08) | 9.51 (9.78)

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Satisfaction Ratings for Both TASK III and ISR Programs Measured by the Caregiver Satisfaction Scale (CSS).
Description: Caregiver satisfaction ratings (usability, ease of use, acceptability) for both TASK III and ISR programs are measured using the Caregiver Satisfaction Scale (CSS). The CSS consists of 9 items rated on a response scale ranging from 1 = Strongly Disagree to 5 = Strongly Agree. Items are summed for a total score, then divided by 9 (number of items) with a possible range of 1 to 5. Higher scores indicate greater satisfaction.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TASK III Group | ISR Group
Number analyzed (Participants) | 31 | 34
score on a scale | 4.59 (.47) | 4.15 (.59)

2. Secondary Outcome: Depressive Symptoms Measured by the Patient Health Questionnaire Depression Scale (PHQ-9).
Description: Caregiver depressive symptoms are measured by the Patient Health Questionnaire Depression Scale (PHQ-9) consisting of 9 items rated on a response scale ranging from 0 = Not at all to 3 = Nearly every day. Items are summed for a total score with a possible range of 0 to 27. Higher scores indicate higher depressive symptoms.
Time Frame: Assessed at Baseline, Week 8, and Week 12, change from Baseline to Week 8 Reported.
Population: As in our prior studies, the number of minutes on the TASK III and ISR calls from the nurse were controlled in our analyses showing data trends as change scores. At each follow-up time point, 8 and 12 weeks, we computed mean differences and 95% CI between groups to evaluate trends in outcomes. Reported here are mean (SE) in change scores from Baseline to 8 weeks.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | TASK III Group | ISR Group
Number analyzed (Participants) | 31 | 34
units on a scale | -2.3 (0.7) | -0.6 (0.7)

3. Secondary Outcome: Life Changes (i.e., Changes in Social Functioning, Subjective Well-being, and Physical Health as a Result of Providing Care) Measured by the Bakas Caregiving Outcomes Scale (BCOS).
Description: Caregiver life changes (i.e., changes in social functioning, subjective well-being, and physical health as a result of providing care) are measured by the Bakas Caregiving Outcomes Scale (BCOS). The BCOS consists of 15 items rated on a response scale ranging from -3 (changed for the worst) to +3 (Changed for the best). The items are recoded (-3 = 1) (-2 = 2) (-1 = 3) (0 = 4) (1 = 5) (2 = 6) (3 = 7) so that positive numbers can be obtained for analysis. The recoded responses to the 15 items are summed for a total score with a possible range of 15-105. Higher scores indicate more positive life changes as a result of providing care.
Time Frame: Assessed at Baseline, Week 8, and Week 12, change from Baseline to Week 8 Reported.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | TASK III Group | ISR Group
Number analyzed (Participants) | 31 | 34
units on a scale | 11.2 (2.6) | 3.1 (2.4)

4. Secondary Outcome: Unhealthy Days Measured by the Number of Unhealthy Days in the Past 30 Days.
Description: Caregiver unhealthy days are measured using the Unhealthy Days (UD) measure consisting of two items: How many days during the past 30 days was your physical health not good?; How many days during the past 30 days was your mental health not good? These items range from 0 = no unhealthy days to 30 = 30 unhealthy days. The two items are summed for a total score, with a cap of 30 days. Higher scores indicate more unhealthy days in the past 30 days.
Time Frame: Assessed at Baseline, Week 8, and Week 12, change from Baseline to Week 8 Reported.
Population: At each follow-up time point, 8 and 12 weeks, we computed mean differences and 95% CI between groups to evaluate trends in outcomes. Reported here are mean (SE) in change scores from Baseline to 8 weeks.
Measure: Mean (Standard Error); unit: Days
Arm/Group | TASK III Group | ISR Group
Number analyzed (Participants) | 31 | 34
Days | 1.93 (1.70) | -1.15 (1.72)

ADVERSE EVENTS:
Time Frame: From Baseline to Week 8 and Week 12.
Description: The clinicaltrials.gov definitions were used.
Arm/Group | TASK III Group | ISR Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT03635151/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT03635151/ICF_001.pdf